CLINICAL TRIAL: NCT03679039
Title: A Single-centre, Prospective, Cohort Trial of the Detection of 5-hydroxymethylcytosine (5-hmC) in Plasma Cell-free DNA for Establishing a Model for Predicting the Efficacy of Conversion Therapy for Patients With Unresectable Colorectal Cancer Liver Metastases
Brief Title: A Model for Predicting the Efficacy of Conversion Therapy for Patients With Colorectal Cancer Liver Metastases by the Detection of 5-hydroxymethylcytosine (5-hmC) in Plasma Cell-free DNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Other Study IDs: PROVE
Record Dates: First submitted 2018-07-16; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Cancer With Liver Metastases
Keywords: colorectal cancer; liver metastases; conversion therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators establish a model for predicting the efficacy of conversion therapy for the patients with unresectable liver metastases of colorectal cancer based on the detection of 5-hydroxymethylcytosine (5-hmC) in training group and validate the effectiveness of the model using a validation group.

DETAILED DESCRIPTION:
Radical resection is the preferred treatment of colorectal cancer patients with liver metastasas which significantly reduce the survival. However, the majority of the patients cannot receive liver lesions resection resulting from the size, number and bad location. Conversion therapy can improve the resection rate of these patients. Unfortunately, the efficacy of conversion therapy is still poor in part of the patients. So, it is crucial to distinguish the beneficial ones from the others.

The aim of this single center study is to establish a model for predicting the efficacy of conversion therapy for the patients with unresectable liver metastases of colorectal cancer based on the detection of 5-hmC. Patients will be eligible for inclusion if they suffer with unresectable liver metastases of colorectal cancer and have not received any anti-tumor treatment. Eligible patients will be assigned to effective group (group A) and drug resistance group (group B) according to the evaluation results of multidisciplinary team after 4-8 cycles of conversion therapy about 2-4 months.

Then, 5-hmC in plasma cell-free DNA will be detected and compared between the two groups of patients (training group) to establish a model to predict the efficacy of convertion therapy of other individuals (validation group) who suffer with unresectable liver metastases of colorectal cancer receiving conversion therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma
* Liver metastases were observed by abdominal pelvic CT and / or MRI with/without other distant metastases
* The liver metastases assessed as unresectable lesions by multidisciplinary team
* No other malignancies in medical history
* Eastern cooperative oncology group score 0-2
* Informed consent

Exclusion Criteria:

* Patients received chemoradiotherapy or other anti-tumor therapy before being enrolled
* Patients and/or family members can not understand or accept this study
* Familial Adenomatous Polyposis, Lynch Syndrome, acute inflammatory bowel disease
* Pregnancy or lactation
* Unsuitable to take part in the clinical trial judged by doctors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable liver metastases from colorectal cancer were not received any anti-tumor therapy before being enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-20 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of the model to predict the drug resistance | 4 months
  Sensitivity and specificity of the model in predicting the drug resistance in conversion therapy for colorectal cancer with unresectable liver metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China